CLINICAL TRIAL: NCT04210362
Title: External Evaluation of the Neurological and Psycho-affective Early Childhood Development Program of the Mexican Non-governmental Organization Un Kilo de Ayuda
Brief Title: External Evaluation of the Neurological and Psycho-affective Early Childhood Development Program of the Mexican NGO Un Kilo de Ayuda
Acronym: NPECDP-UKA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to the Covid-19 contingency, activities were suspended in March 2020. Baseline measurements were obtained for n=764 children whose caregivers enrolled in the NPECDP-UKA.
Sponsor: Amado David Quezada Sánchez (Other Government)
Collaborators: Un Kilo de Ayuda A.C. (Unknown); Instituto Nacional de Perinatologia Isidro Espinosa de los Reyes (Other Government)
Responsible Party: Sponsor-Investigator, Amado David Quezada Sánchez, Reseracher in Medical Sciences, Mexican National Institute of Public Health
Organization: Mexican National Institute of Public Health (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1538/CI-896-2018/CB18-317
Record Dates: First submitted 2019-07-14; First posted 2019-12-24 (Actual); Last update posted 2022-08-25 (Actual); Status verified 2022-08

CONDITIONS: Child Development
Keywords: neurodevelopment; responsive caregiving; nuturing care; counseling

STUDY DESIGN:
Intervention Model Description: A variation of the stepped wedge cluster randomized trial design was specified. Due to ethical and logistical considerations, the intervention in study groups under this design starts sequentially but measurements are performed at the same time period in all groups. The key difference between groups is thus the time of exposure to the intervention. Clusters were randomized into four study groups (30, 24, and 12 months of exposure, and a non-exposed group). The intervention consists of educational workshops for caregivers aimed at promoting healthy nurturing care practices and responsive caregiving. Assessment of intervention effects is performed as in a parallel design.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Educational intervention for 30 months (Experimental): Children aged 31 to 60 months and their caregivers from 20 municipalities of Oaxaca will have been exposed to the Neurobehavioral and Psycho-affective Development Program for 30 months.
  Interventions: Behavioral: Workshops on responsive caregiving
- Educational intervention for 24 months (Experimental): Children aged 31 to 60 months and their caregivers from 20 municipalities of Oaxaca will have been exposed to the Neurobehavioral and Psycho-affective Development Program for 24 months.
  Interventions: Behavioral: Workshops on responsive caregiving
- Educational intervention for 12 months (Experimental): Children aged 31 to 60 months and their caregivers from 20 municipalities of Oaxaca will have been exposed to the Neurobehavioral and Psycho-affective Development Program for 12 months.
  Interventions: Behavioral: Workshops on responsive caregiving
- Comparison group (No Intervention): Group comprised of children aged 31 to 60 months and their caregivers from 20 municipalities of Oaxaca, Mexico. Children and their caregivers will not be exposed to the intervention at the moment of their measurements.

INTERVENTIONS:
Behavioral: Workshops on responsive caregiving — Caregivers will receive monthly workshops about several dimensions of nurturing care, responsive caregiving and early child development. Workshops will be reinforced through home visits.
  Arms: Educational intervention for 12 months; Educational intervention for 24 months; Educational intervention for 30 months

SUMMARY:
Investing in early childhood development is one of the best cost-effective investments a country can make to boost long term economic growth, promote peaceful and sustainable societies, contribute to tackle poverty traps and eradicate inequality. It is also necessary to uphold the right of every child to survive and thrive. The single most powerful context for nurturing care is the immediate home, often mainly provided by mothers.

Although the Mexican government has implemented social programs in the past, some with nutrition and child development components, poor and isolated communities have not benefited as others easier to reach. This is particularly true for the State of Oaxaca given its orography, where higher levels of malnutrition and a higher risk of suboptimal neurodevelopment are present.

Since 1989, Un Kilo de Ayuda A.C. (UKA), a nongovernmental organization, has been involved in preventing child undernutrition in contexts of high poverty. Currently, UKA has 9 Early Childhood Development Centers distributed in 5 States of Mexico, including Oaxaca. UKA has developed the Neurological and Psycho-affective Early Childhood Development Program (NPECDP-UKA) that seeks to contribute to timely stimulation in children under 5 years of age and promote perceptual parenting practices. As part of the NPECDP-UKA, UKA redesigned their interventions to promote healthy nurturing care practices and responsive caregiving through workshops provided to caregivers and pregnant women, and with reinforcement through home visits.

It is in the interest of this study to evaluate the NPECDP-UKA through a variation of a stepped wedge cluster randomized trial. The study sample consists of participants from 80 municipalities of Oaxaca (~50% with high or very high margination status), 20 municipalities were randomly assigned to each arm. Study arms differ by design on the time of exposure to the program (0,18,24 and 30 months at the final measurement). Subjects from all study groups share the characteristic to be enrolled in the NPECDP-UKA, the group with 0 months of exposure will serve as a comparison group. This distinctive characteristic of the study requires a progressive incorporation of study groups to be able to compare development measurements between study groups at the same ages and among subjects all enrolled in the program to avoid self-selection bias. The main study hypothesis states that children exposed to the Program will have better neurodevelopment outcomes than those not exposed.

This study will provide evidence of the effect of an educational intervention for caregivers on the neurodevelopment of children under 5 years of age. Currently evidence of such interventions is very limited, especially for interventions performed by a nongovernmental organization. This is the first evaluation of this kind in Mexico.

ELIGIBILITY:
Inclusion Criteria

* Communities: Municipalities in the State of Oaxaca where the NPECDP-UKA is not currently operating.
* Whithin selected communities:

children aged1 to 60 months and their caregivers who decided to enroll in the NPECDP-UKA.

Exclusion Criteria (communities):

* Communities: Municipalities in the State of Oaxaca with a population of children under 5 years of age below 35 habitants according to the Census of 2010

Ages: 1 Month to 60 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 764 (Actual)
Dates: Start 2019-07-15 (Actual); Primary Completion 2020-02-10 (Actual); Study Completion 2020-02-10 (Actual)

PRIMARY OUTCOMES:
Child Development Evaluation Test 2nd Edition (CDE-II) | Up to 30 months
  The CDE-II, or Evaluación del Desarrollo Infantil (EDI-II) in Spanish, was developed and validated in Mexico to screen populations for lag and for risk of delay in child development. The test has specific items for 14 age groups of children aged 1 to 60 months. Assessed developmental areas include gross motor skills, fine motor skills, language, social skills, and cognitive skills. The CDE-II is based on age-group specific items, score results are categorized into three levels: Green (normal development), Yellow (developmental lag) and Red (at risk of development delay)

SECONDARY OUTCOMES:
Verbal McCarthy Scale of Children's Abilities (MSCA) | Up to 30 months
  The verbal MSCA has an arbitrarily chosen mean of 50 and stadard deviation of 10. Higher values indicate a higher level of the measured dimension.
Perceptual-performance McCarthy Scale of Children's Abilities (MSCA) | Up to 30 months
  The perceptual-performance MSCA has an arbitrarily chosen mean of 50 and stadard deviation of 10. Higher values indicate a higher level of the measured dimension.
Quantitative McCarthy Scale of Children's Abilities (MSCA) | Up to 30 months
  The quantitative MSCA has an arbitrarily chosen mean of 50 and stadard deviation of 10. Higher values indicate a higher level of the measured dimension.
Memory McCarthy Scale of Children's Abilities (MSCA) | Up to 30 months
  The memory MSCA has an arbitrarily chosen mean of 50 and stadard deviation of 10. Higher values indicate a higher level of the measured dimension.
Motor McCarthy Scale of Children's Abilities (MSCA) | Up to 30 months
  The motor MSCA has an arbitrarily chosen mean of 50 and stadard deviation of 10. Higher values indicate a higher level of the measured dimension.
General Cognitive Index from McCarthy Scales of Children's Abilities (MSCA) | Up to 30 months
  The General Cognitive Scale is obtained adding up the verbal, percetual-performance and quantitative MSCA and it is converted into the General Cognitive Index (GCI). The GCI has a mean set at 100 and a standard deviation of 16.

CONTACTS AND LOCATIONS:
Overall Officials: Edson Serván-Mori, PhD, Principal Investigator — Mexican National Institute of Public Health
Locations (1):
- Un Kilo de Ayuda, A.C., Oaxaca City, Mexico

REFERENCES:
- [Background] Van der Gaag J, Tan J-P. The benefits of early child development programs: an economic analysis. World Bank Group; 1998
- [Background] Heckman JJ, Moon SH, Pinto R, Savelyev P, Yavitz A. A new cost-benefit and rate of return analysis for the Perry Preschool Program: A summary. Cambridge, MA 02138: National Bureau of Economic Research; 2010. (NBER Working Paper). Report No.: 16180
- [Background] Heckman J, Carneiro P. Human capital policy. Cambridge, MA 02138: National Bureau of Economic Research; 2003. (NBER Working Paper). Report No.: 9495
- [Background] Delalibera BR, Ferreira PC. Early childhood education and economic growth. J Econ Dyn Control. 2019;98:82-104
- [Background] Organization WH, Fund UNC, Group WB. Nurturing care for early childhood development: a framework for helping children survive and thrive to transform health and human potential. Ginebra 27, Suiza: World Health Organization; 2018
- [Background] Bick J, Nelson CA. Early Adverse Experiences and the Developing Brain. Neuropsychopharmacology. 2016 Jan;41(1):177-96. doi: 10.1038/npp.2015.252. Epub 2015 Sep 3. PMID 26334107
- [Background] Shonkoff JP, Garner AS; Committee on Psychosocial Aspects of Child and Family Health; Committee on Early Childhood, Adoption, and Dependent Care; Section on Developmental and Behavioral Pediatrics. The lifelong effects of early childhood adversity and toxic stress. Pediatrics. 2012 Jan;129(1):e232-46. doi: 10.1542/peds.2011-2663. Epub 2011 Dec 26. PMID 22201156
- [Background] Force LMT. Toward Universal Learning: What Every Child Should Learn. Washington/Montreal: Brookings/UIS. 2013
- [Background] Child C on the D. The Science of Early Childhood Development Closing the Gap Between What We Know and What We Do [Internet]. Cambridge, MA 02138; 2007. Available from: https://developingchild.harvard.edu/wp-content/uploads/2015/05/Science_Early_Childhood_Development.pdf
- [Background] Duncan GJ, Dowsett CJ, Claessens A, Magnuson K, Huston AC, Klebanov P, Pagani LS, Feinstein L, Engel M, Brooks-Gunn J, Sexton H, Duckworth K, Japel C. School readiness and later achievement. Dev Psychol. 2007 Nov;43(6):1428-1446. doi: 10.1037/0012-1649.43.6.1428. PMID 18020822
- [Background] Blair C, Razza RP. Relating effortful control, executive function, and false belief understanding to emerging math and literacy ability in kindergarten. Child Dev. 2007 Mar-Apr;78(2):647-63. doi: 10.1111/j.1467-8624.2007.01019.x. PMID 17381795
- [Background] Shonkoff JP, Boyce WT, McEwen BS. Neuroscience, molecular biology, and the childhood roots of health disparities: building a new framework for health promotion and disease prevention. JAMA. 2009 Jun 3;301(21):2252-9. doi: 10.1001/jama.2009.754. PMID 19491187
- [Background] Caspi A, Moffitt TE, Newman DL, Silva PA. Behavioral observations at age 3 years predict adult psychiatric disorders. Longitudinal evidence from a birth cohort. Arch Gen Psychiatry. 1996 Nov;53(11):1033-9. doi: 10.1001/archpsyc.1996.01830110071009. PMID 8911226
- [Background] Heckman JJ. Skill formation and the economics of investing in disadvantaged children. Science. 2006 Jun 30;312(5782):1900-2. doi: 10.1126/science.1128898. PMID 16809525
- [Background] Young ME. Addressing and mitigating vulnerability across the life cycle: The case for investing in early childhood. UNDP Hum Dev Rep Off. 2014
- [Background] The United Natons Children's Fund (UNICEF). The 2030 Agenda for Sustainable Development [Internet]. UNICEF and the SDGs. 2016. Available from: https://www.unicef.org/agenda2030/69525.html
- [Background] Britto PR, Lye SJ, Proulx K, Yousafzai AK, Matthews SG, Vaivada T, Perez-Escamilla R, Rao N, Ip P, Fernald LCH, MacMillan H, Hanson M, Wachs TD, Yao H, Yoshikawa H, Cerezo A, Leckman JF, Bhutta ZA; Early Childhood Development Interventions Review Group, for the Lancet Early Childhood Development Series Steering Committee. Nurturing care: promoting early childhood development. Lancet. 2017 Jan 7;389(10064):91-102. doi: 10.1016/S0140-6736(16)31390-3. Epub 2016 Oct 4. PMID 27717615
- [Background] National Research Council (US) and Institute of Medicine (US) Committee on Integrating the Science of Early Childhood Development; Shonkoff JP, Phillips DA, editors. From Neurons to Neighborhoods: The Science of Early Childhood Development. Washington (DC): National Academies Press (US); 2000. Available from http://www.ncbi.nlm.nih.gov/books/NBK225557/ PMID 25077268
- [Background] Britto PR, Engle P. Parenting education and support: maximizing the most critical enabling environment. In: Marope P, Kaga Y, editors. Investing against evidence: the global state of early childhood care and education. 1st ed. Paris, France; 2015. p. 157.
- [Background] Consejo Nacional de Evaluación de la Política de Desarrollo Social (CONEVAL). Estadísticas de pobreza en Oaxaca [Internet]. Información de Pobreza y Evaluación de las Entidades Federativa. Available from: https://www.coneval.org.mx/coordinacion/entidades/Oaxaca/Paginas/principal.aspx
- [Background] Hemming K, Haines TP, Chilton PJ, Girling AJ, Lilford RJ. The stepped wedge cluster randomised trial: rationale, design, analysis, and reporting. BMJ. 2015 Feb 6;350:h391. doi: 10.1136/bmj.h391. No abstract available. PMID 25662947
- [Background] McCarthy D. McCarthy Scales of Childrens Abilities. New York: The Psychological Corporation. 1972.
- [Derived] Servan-Mori E, Quezada-Sanchez AD, Fuentes-Rivera E, Pineda-Antunez C, Hernandez-Chavez MDC, Garcia-Martinez A, Garcia-Feregrino R, Madrigal A, Guerrero B, Medrano G, Schnaas L. Proximal determinants of suboptimal early child development during the first three years of life in socially deprived Mexican contexts. PLoS One. 2023 Nov 2;18(11):e0291300. doi: 10.1371/journal.pone.0291300. eCollection 2023. PMID 37917638
- [Derived] Servan-Mori E, Fuentes-Rivera E, Quezada AD, Pineda-Antunez C, Del Carmen Hernandez-Chavez M, Garcia-Martinez A, Madrigal A, Garcia-Feregrino R, Santiago-Angelino T, Hernandez-Serrato M, Schnaas L. Early neurological development and nutritional status in Mexican socially deprived contexts. PLoS One. 2022 Jun 21;17(6):e0270085. doi: 10.1371/journal.pone.0270085. eCollection 2022. PMID 35727758
- [Derived] Quezada-Sanchez AD, Fuentes-Rivera E, Garcia-Martinez A, Del Carmen Hernandez-Chavez M, Pineda-Antunez C, Martinez MR, Garcia-Guerra A, Garcia-Feregrino R, Madrigal-Ramirez A, Santiago-Angelino T, Olvera-Flores F, Schnaas L, Perez-Escamilla R, Servan-Mori E. Assessing the effect of an educational intervention on early childhood development among Mexican preschool children in the state of Oaxaca: a study protocol of a cluster randomized stepped-wedge trial. Trials. 2022 Feb 8;23(1):126. doi: 10.1186/s13063-022-06024-2. PMID 35130939